CLINICAL TRIAL: NCT06745193
Title: A Prospective, Randomized, Open, Phase II Clinical Study of Chidamide in Combination with Camrelizumab and Apatinib for Advanced Esophageal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-Q73
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Advanced Esophageal Carcinoma
MeSH Terms: interventions — Irinotecan; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- chidamide+Camrelizumab+Apatinib (Experimental)
  Interventions: Drug: chidamide+Camrelizumab+Apatinib
- SOC (Placebo Comparator): Irinotecan or Docetaxel or Paclitaxel
  Interventions: Drug: Irinotecan or Docetaxel or Paclitaxel

INTERVENTIONS:
Drug: chidamide+Camrelizumab+Apatinib — chidamide+Camrelizumab+Apatinib
  Arms: chidamide+Camrelizumab+Apatinib
Drug: Irinotecan or Docetaxel or Paclitaxel — Irinotecan Docetaxel Paclitaxel
  Arms: SOC

SUMMARY:
This study aims to evaluate the efficacy and safety of a combination treatment of chidamide, camrelizumab, and apatinib in patients with advanced esophageal cancer. This open-label, phase II clinical trial will involve randomly assigning participants to receive either the combination of these drugs or a standard treatment. The primary endpoints is ORR and the second endpoints include progression-free survival and overall survival, while safety will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

- Age ≥ 18 years and ≤ 75 years, regardless of gender; Histologically or cytologically confirmed locally advanced/metastatic esophageal squamous cell carcinoma; A total of 1-3 lines of prior treatment for advanced disease; If prior immunotherapy has been used, the duration of single-line immunotherapy must be greater than 6 months; ECOG performance status of 0-1; At least one measurable lesion (according to RECIST v1.1 assessment criteria); Absolute neutrophil count ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 90 g/L;

Functionality requirements for other organs must be met:

Cardiac function: Left ventricular ejection fraction ≥ 50%, no organic arrhythmias; Liver function: ALT and AST ≤ 2.5 times the upper limit of normal (if with liver metastases, ALT and AST ≤ 5 times the upper limit of normal), total bilirubin ≤ 1.5 times the upper limit of normal; Kidney function: Creatinine ≤ 1.5 times the upper limit of normal; Coagulation function: International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal; Prothrombin Time (PT) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times the upper limit of normal (unless the subject is receiving anticoagulant treatment and PT and APTT are within the expected range for those on anticoagulant therapy during screening); Thyroid function: Thyroid Stimulating Hormone (TSH) or free Thyroxine (FT4) or free Triiodothyronine (FT3) should all be within ±10% of normal range.

Expected survival time ≥ 3 months; Non-surgically sterilized or women of childbearing potential must use a medically recognized contraceptive method (such as an intrauterine device, contraceptive pills, or condoms) during the study treatment period and for 3 months after the end of the study treatment; non-surgically sterilized women of childbearing potential must have a negative serum or urine HCG test within 72 hours prior to enrollment; they must also not be breastfeeding; male patients with partners who are women of childbearing potential should use effective contraception during the trial and for 3 months after the last administration.

Participants must voluntarily agree to participate in this clinical trial and sign a written informed consent form.

Exclusion Criteria:

- Previous treatment with HDAC inhibitors or anti-angiogenic agents; Symptomatic or active progression of central nervous system (CNS) metastases; The patient has any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; patients with vitiligo; childhood asthma that has completely resolved and requires no intervention in adulthood may be included; patients with asthma requiring bronchodilators for medical intervention cannot be included); The patient is currently using immunosuppressants or systemic corticosteroids for immunosuppressive purposes (dosage > 10 mg/day of prednisone or other equivalent corticosteroids) and has continued use in the 2 weeks prior to enrollment; Presence of active infection requiring systemic treatment; History of severe allergic reactions to other monoclonal antibodies; Uncontrolled clinical symptoms or diseases of the heart, such as: NYHA class II heart failure or above; unstable angina; myocardial infarction within the past year; clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention; QTc interval prolonged to > 480 ms; Presence of bleeding tendencies or currently undergoing thrombolysis or anticoagulant treatment; preventive use of low-dose aspirin or low molecular weight heparin is permitted; Significant clinically meaningful hemorrhagic symptoms or clear bleeding tendencies within 3 months prior to enrollment, such as hemoptysis of 2.5 ml or more, gastrointestinal bleeding, esophageal-cardiac varices at risk of bleeding, hemorrhagic gastric ulcers, or vasculitis; Occurrence of arterial/venous thromboembolism events within 6 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, intracerebral hemorrhage, cerebral infarction), deep venous thrombosis, or pulmonary embolism; Known hereditary or acquired bleeding and thrombotic tendencies (e.g., hemophiliacs, coagulation disorders, thrombocytopenia, etc.); Presence of hypertension that cannot be adequately controlled by antihypertensive medication (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg); Urinalysis indicates urine protein ≥ ++ and confirmed 24-hour urine protein amount > 1.0 g; Patients who have previously received radiotherapy, chemotherapy, hormone therapy, or surgery, with less than 4 weeks since treatment completion (last dose) before the study medication; patients who have undergone molecular targeted therapy (including other oral targeted drugs in clinical trials) within less than 5 half-lives of the medication prior to the first dose of study medication, or patients who have not recovered from adverse events (except alopecia) to ≤ CTCAE grade 1; Severe local invasion of lesions with risks of organ leakage, significant hemorrhage, or perforation; Known presence of other malignant tumors that are currently progressing or require active treatment; Patients participating in other clinical trials; HIV positive; HCV positive; HBsAg or HBcAb positive with concurrent detection of positive HBV DNA copy number (quantitative detection limit of 500 IU/ml); Administration of live vaccines within 4 weeks prior to the start of treatment; Based on the investigator's judgment, other severe, acute, or chronic medical conditions, mental disorders, or laboratory abnormalities that may increase the risks associated with participation in the study or may interfere with the interpretation of study results may also exclude the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | up to 24 months

SECONDARY OUTCOMES:
progression free surival（PFS） | up to 24 months
overall surival（OS） | up to 24 months
Adverse events | up to 24 months
Disease Control Rate（DCR） | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China